CLINICAL TRIAL: NCT01280422
Title: Analysis of Drug-drug Interaction Alert Based on Multicenter Clinical Database
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Yu-Chuan Li, Department of Dermatology, WanFang Hospital
Other Study IDs: 99009
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Drug Interaction Alert
Keywords: ROCDR

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The doctor's overridden rate for Drug-drug interaction (DDI) alert systems was 85-95% in foreign and there was more than 90% overridden rate in Taiwan. Why DDI alerts systems which spent much time and money to establish could not use medicinal information to increase drug safety? One of the reasons which induced to override was that health care thought there were too much DDI alerts and high false alerts.

The difference between DDI alert systems from pharmacists to confirm drug-drug interaction was that pharmacists not only confirmed ordering drug at the same time but also checked the other drug information such as frequency, rote and refill etc. Therefore, DDI alert systems which were established by drug code alone would induce a lot of false alerts.

In order to study how much false alert rate in drug-drug interactions, this research selected most common drug-drug interaction which was antacids and antibiotics. Antacids were most self-payment so this research needed to analyze ROCDR (Establishing a Multi-Center, Longitudinal, Research-Oriented Clinical Data Repository for Clinical Research). The aim was to study how many drug-drug interactions and false alerts from antacids and antibiotics and analyze the difference in different department. Finally, proposing advice and assessment for building drug-drug interaction alerts system to strength drug information system and increase drug safety.

ELIGIBILITY:
Inclusion Criteria:

* Select DDI rules: antacids and antibiotics
* Database: ROCDR (multicenter clinical database)
* The pharmacists defined six rules which were based on medical knowledge for true alerts or false-alert.

  1. True alert: Rule 1 and Rule 2
  2. "False-alert": Rule 3 or Rule 4
  3. "Other" (Unable to determine): Rule 5 or Rule 6

Exclusion Criteria:

* N/A

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 67128927 (Actual)
Dates: Start 2010-02; Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan Li, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan